CLINICAL TRIAL: NCT01954472
Title: The Effect of an Enhanced Dietary Portfolio Plus Exercise on Cardiovascular Risk in High Risk Individuals.
Brief Title: Enhanced Multicenter Dietary Portfolio Study
Acronym: EDP8
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was combined with another CIHR funded study (NCT02078635). Both studies involve the same dietary portfolio and the same study population.
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other); Laval University (Other); University of Manitoba (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 13-188; FRN 130278 (Other Grant/Funding Number: Canadian Institutes of Health Research, Operating Grant)
Record Dates: First submitted 2013-09-23; First posted 2013-10-01 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases; Type 2 Diabetes; Hypercholesterolemia
Keywords: Portfolio diet; dietary modification; hypercholesterolemia; diabetes; Exercise; CVD risk; glycemic index; inflammatory biomarkers; monounsaturated fat; saturated fat; nuts; plant sterols; vegetable protein; viscous fiber; soy
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Hypercholesterolemia; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Portfolio plus structured exercise (Experimental): Diet: The dietary portfolio advice: to limit saturated fat to <7% of total calories and cholesterol to <200 mg/d) plus inclusion of viscous fibres, soy protein, plant sterols and nuts, 5% extra monounsaturated fat, and selection of low glycemic index foods and will emphasize current recommendations for fruit and vegetable intakes (5-10 servings/d).
  Interventions: Behavioral: Enhanced portfolio plus structured exercise
- High fiber diet plus routine exercise (Active Comparator): A diet of whole grain foods (brown rice, whole wheat breads, muffins and breakfast cereals); reduced meat consumption; lower fat dairy foods and a control margarine
  Interventions: Behavioral: High fiber diet plus routine exercise

INTERVENTIONS:
Behavioral: Enhanced portfolio plus structured exercise — Foods on the dietary portfolio plan will contribute 9g/1000 kcal viscous fibre as β-glucan (oats, barley, oat bran breads and soups) and psyllium (cereal), 1g plant sterol/1000 kcal diet (in sterol margarine), 22.5g soy protein/1000 kcal (soy burgers, dogs, links, other soy meat analogues, soy milks, yogurts and cheese), and additional sources of plant protein from pulses (eg. Lentils, chickpeas, beans, etc) and 22.5g almonds or equivalent of other nuts/1000 kcal and increased MUFA (as olive and canola oils, avocados, nuts, margarine and salad dressings). The glycemic index will be reduced from 83 to 70 GI units (bread scale).
  Exercise: The physical activity/exercise program is based on the program used at the Quebec Heart and Lung Institute.
  Other Names: Dietary Portfolio of cholesterol-lowering foods; Laval exercise program
  Arms: Enhanced Portfolio plus structured exercise
Behavioral: High fiber diet plus routine exercise — Dietary advice will be given to encourage intake of whole grain foods (brown rice, whole wheat breads, muffins and breakfast cereals); to reduce meat consumption, choose low fat dairy products and a control margarine.
  Exercise: A pamphlet (Canada's Physical Activity Guide, Health Canada) encouraging increased physical activity will be provided.
  Arms: High fiber diet plus routine exercise

SUMMARY:
"Is it possible to recruit and retain up to 200 participants in a Randomize Control Trial (RCT) of high impact lifestyle approach of diet and exercise designed to significantly reduce cardiovascular events in middle-aged and older men and women at high risk of such events?" To address this question, we propose a pilot study of 3 years in duration: 1 year recruitment and randomization, a full year of intervention for all recruited participants, and the last 6 months to assess the one year data and prepare and submit the full trial application, informed by the pilot study outcomes in terms of retention rate. The pilot will then continue on for the full 9 years of intervention and be rolled into the main study involving additional Canadian centers and collaborating international centers in the US, Britain, Europe, Australia, New Zealand, India, and South Africa.

DETAILED DESCRIPTION:
There is a major need for a large RCT to demonstrate the effect of lifestyle modification (diet and exercise) on cardiovascular disease (CVD) outcomes. The pilot study will demonstrate the feasibility as a prerequisite for continuing on to the large RCT. Large RCT: This trial will test the effect of a high impact dietary approach combining foods with functional effects, including LDL-cholesterol (LDL-C) and blood pressure (BP) reduction, together with an exercise program which has been associated with reduction in carotid atheroma assessed by MRI. The combined approach will have a more significant effect on CVD risk factors than previous trials and will be compared with a high cereal fibre diet and exercise advice, consistent with good clinical practice, in a randomized parallel trial of 9 years duration. ~6,000 high risk participants will be recruited comprising individuals with 1) type 2 diabetes, 2) post myocardial infarction (MI), and 3) Statin intolerant individuals. The primary outcome will be CVD event (MI, and stroke, fatal and non-fatal) (1). We believe we will achieve a 20% reduction in CVD events with ~10% related to diet reflected in reduction in traditional risk factors (LDL-C, BP) and 10% to exercise and increased cardiovascular fitness at year 9.

Pilot Study: We therefore propose to undertake a 1 year pilot study with 200 participants to demonstrate feasibility: 1) Successful recruitment (200 participants/year) and 2) retention (>90%)

Background: We have demonstrated the specific CVD reducing potential of the proposed components of our dietary intervention in a series of CIHR funded studies. The core dietary components (dietary portfolio of FDA approved cholesterol-lowering foods) in our recent CIHR-funded trial reduced LDL-C by 13-14% (JAMA 2011) with reductions also in diastolic blood pressure over 6 months. The CVD risk score was reduced by ~10% on the treatment. This approach will be combined with increased levels of monounsaturated fat (MUFA) which in a further CIHR-funded portfolio study raised HDL-C and reduced the total:HDL-C ratio (CMAJ 2010) resulting in an ~11% CVD risk score reduction on the high MUFA compared to the low MUFA portfolio. Low glycemic index foods will be selected which in our CIHR-funded trial in type 2 diabetes increased HDL-C and reduced HbA1c, the total:HDL-C ratio (JAMA 2008) and, with the added emphasis on legumes (dried peas, beans, lentils), significantly reduced BP leading to a CVD risk score reduction of ~5% (Arch Intern Med 2012). We consider this dietary package to have major potential in CVD risk reduction with a possible reduction in relative risk of 24% in the absence of negative or positive interactions.

The physical activity/exercise intervention is the end-product of a 25 year cumulative experience of investigators of the Quebec Heart and Lung Institute regarding physical activity/exercise prescriptions to various types of individuals/patients. Our program has also been recently tested in high risk patients with documented coronary artery disease managed by coronary artery bypass graft procedure (with/without type 2 diabetes). Unpublished preliminary results from this latter intervention in high risk patients indicate that our program not only induces substantial improvements in the CVD risk factor profile beyond clinical guidelines-aligned with optimal pharmacotherapy but that such an intervention appears to induce a significant reduction in carotid artery atherosclerosis assessed by magnetic resonance imaging. The latest meta-analysis estimated that only 150 min/week of moderate exercise reduced CHD risk by 14%. Our Laval program with a 420 min/wk of moderate exercise plus additional structured exercise would therefore also reduce CVD risk by at least 14% (or as much as 39% if the relationship between exercise time and CVD risk reduction were linear). The program aims to reduce sedentary behavior. It is safe and affordable in clinical practice. At a cost of about $900 per patient in the first year where the major training takes place, it is considerably less expensive than the DPP, DPS and Look AHEAD trials.

The research questions are therefore:

1. What is the feasibility in terms of recruitment and retention of implementing a high impact diet and physical activity/exercise program for CVD prevention in high risk or statin-intolerant individuals?
2. Based on the observed retention in the pilot study, the required recruitment for the large trial can be refined, if necessary.

ELIGIBILITY:
A) Inclusion Criteria:

Eligible participants will be:

1. men, over 50
2. postmenopausal women, over 60 or
3. postmenopausal women under 60 with a family history of hypercholesterolemia and 1 CVD risk factor.

Participants will have the following characteristics:

* BMI 25-40 kg/m2 with body weight that has remained constant (within ±3%) over the last 3 months preceding the onset of the study
* Plus at least 1 of the following 3 criteria:

  1. have type 2 diabetes with one of the following:

     * raised LDL-C(in accordance with the 2012 Canadian Cardiovascular Society Guidelines)
     * raised BP (> 130/80mmHg), or
     * active smoking;
  2. be non-diabetic subjects post MI or post percutaneous coronary intervention (angioplasty) on statin therapy; and
  3. have a modified Framingham risk score >20% (CCS 2012) and are unable (intolerant) or unwilling to take statin drugs.

B) Exclusion Criteria:

Individuals with the following conditions will be excluded:

* cardiovascular disease that precludes exercise e.g.

  * recent stroke or
  * myocardial infarction, or
* cardiac condition that compromises normal function

  * mitral valve disease,
  * heart failure--grades 2-4 (New York Heart Association classification),
  * severe angina or
  * other conditions preventing exercise,
* secondary causes of hypercholesterolemia

  * hypothyroidism, (unless treated and on a stable dose of L-thyroxine)
  * renal or liver disease
* uncontrolled blood pressure
* major disability
* disorder requiring continuous medical attention and treatment:

  * chronic heart failure,
  * liver disease,
  * renal failure or
  * cancer (except non-melanoma skin cancer--basal cell, squamous cell),
* chronic infections (bacterial or viral)
* chronic inflammatory diseases (e.g. lupus, ulcerative colitis)
* other autoimmune diseases
* major surgery <6 months prior to randomization
* alcohol consumption >2 drinks/d.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-10-07 (Actual); Study Completion 2014-10-07 (Actual)

PRIMARY OUTCOMES:
Feasibility measured by recruitment and retention rates | 1 year in a 9 year study
  Pilot study: Recruitment and retention rates will establish the feasibility of proceeding to the large RCT ie the 9 year intervention study.
  Long term study (9 years intervention): Non-fatal MI, non-fatal stroke and CV mortality as defined by MACE.

SECONDARY OUTCOMES:
Serum lipids: total cholesterol, LDL-chol, HDL-chol and Triglycerides | At months -3, -2, -1 and then at months 0, 3, 6 and 12
C-reactive protein | At months -3, -2, -1 and then at months 0, 3, 6 and 12
Hemoglobin A1c | At months -3, -2, -1 and then at months 0, 3, 6 and 12
Glucose | At months -3, -2, -1 and then at months 0, 3, 6 and 12
Blood Pressure | At months -3, -2, -1 and then at months 0, 3, 6 and 12
treadmill testing | At months 0 and 12
diet history | At months -3, -2, -1 and then at months 0, 3, 6 and12
Pedometer records | At months 0, 2, 4, 6, 8, 10 and 12
Exercise history | At months 0, 3, 6, and 12

CONTACTS AND LOCATIONS:
Overall Officials: David J Jenkins, MD, Principal Investigator — St. Michael's Hospital / University of Toronto; Benoit lamarche, PhD, Study Director — Laval University; Peter Jones, PhD, Study Director — University of Manitoba; Jiri Frohilich, MD, Study Director — University of British Columbia
Locations (4):
- Canada (4):
  - Healthy Heart Lipid Clinic, St. Paul's Hospital, Vancouver, British Columbia
  - Richardson Center for Functional Foods and Nutraceuticals and the St. Boniface Hospital Cardiovascular Center, University of Manitoba, Winnipeg, Manitoba
  - Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario
  - Institute of Nutraceuticals and Functional Foods and the Quebec Heart and Lung Institute, Laval University, Québec, Quebec

REFERENCES:
- [Background] Jenkins DJ, Jones PJ, Lamarche B, Kendall CW, Faulkner D, Cermakova L, Gigleux I, Ramprasath V, de Souza R, Ireland C, Patel D, Srichaikul K, Abdulnour S, Bashyam B, Collier C, Hoshizaki S, Josse RG, Leiter LA, Connelly PW, Frohlich J. Effect of a dietary portfolio of cholesterol-lowering foods given at 2 levels of intensity of dietary advice on serum lipids in hyperlipidemia: a randomized controlled trial. JAMA. 2011 Aug 24;306(8):831-9. doi: 10.1001/jama.2011.1202. PMID 21862744
- [Background] Jenkins DJ, Chiavaroli L, Wong JM, Kendall C, Lewis GF, Vidgen E, Connelly PW, Leiter LA, Josse RG, Lamarche B. Adding monounsaturated fatty acids to a dietary portfolio of cholesterol-lowering foods in hypercholesterolemia. CMAJ. 2010 Dec 14;182(18):1961-7. doi: 10.1503/cmaj.092128. Epub 2010 Nov 1. PMID 21041432
- [Background] Jenkins DJ, Kendall CW, Augustin LS, Mitchell S, Sahye-Pudaruth S, Blanco Mejia S, Chiavaroli L, Mirrahimi A, Ireland C, Bashyam B, Vidgen E, de Souza RJ, Sievenpiper JL, Coveney J, Leiter LA, Josse RG. Effect of legumes as part of a low glycemic index diet on glycemic control and cardiovascular risk factors in type 2 diabetes mellitus: a randomized controlled trial. Arch Intern Med. 2012 Nov 26;172(21):1653-60. doi: 10.1001/2013.jamainternmed.70. PMID 23089999
- [Background] Borel AL, Nazare JA, Smith J, Almeras N, Tremblay A, Bergeron J, Poirier P, Despres JP. Visceral and not subcutaneous abdominal adiposity reduction drives the benefits of a 1-year lifestyle modification program. Obesity (Silver Spring). 2012 Jun;20(6):1223-33. doi: 10.1038/oby.2011.396. Epub 2012 Jan 19. PMID 22262155
- [Background] Borel AL, Nazare JA, Smith J, Almeras N, Tremblay A, Bergeron J, Poirier P, Despres JP. Improvement in insulin sensitivity following a 1-year lifestyle intervention program in viscerally obese men: contribution of abdominal adiposity. Metabolism. 2012 Feb;61(2):262-72. doi: 10.1016/j.metabol.2011.06.024. Epub 2011 Aug 23. PMID 21864868
- [Background] Pelletier-Beaumont E, Arsenault BJ, Almeras N, Bergeron J, Tremblay A, Poirier P, Despres JP. Normalization of visceral adiposity is required to normalize plasma apolipoprotein B levels in response to a healthy eating/physical activity lifestyle modification program in viscerally obese men. Atherosclerosis. 2012 Apr;221(2):577-82. doi: 10.1016/j.atherosclerosis.2012.01.023. Epub 2012 Jan 20. PMID 22321874
- [Background] Jenkins DJ, Kendall CW, McKeown-Eyssen G, Josse RG, Silverberg J, Booth GL, Vidgen E, Josse AR, Nguyen TH, Corrigan S, Banach MS, Ares S, Mitchell S, Emam A, Augustin LS, Parker TL, Leiter LA. Effect of a low-glycemic index or a high-cereal fiber diet on type 2 diabetes: a randomized trial. JAMA. 2008 Dec 17;300(23):2742-53. doi: 10.1001/jama.2008.808. PMID 19088352
- [Background] Jenkins DJ, Kendall CW, Faulkner D, Vidgen E, Trautwein EA, Parker TL, Marchie A, Koumbridis G, Lapsley KG, Josse RG, Leiter LA, Connelly PW. A dietary portfolio approach to cholesterol reduction: combined effects of plant sterols, vegetable proteins, and viscous fibers in hypercholesterolemia. Metabolism. 2002 Dec;51(12):1596-604. doi: 10.1053/meta.2002.35578. PMID 12489074
- [Background] Jenkins DJ, Kendall CW, Faulkner DA, Nguyen T, Kemp T, Marchie A, Wong JM, de Souza R, Emam A, Vidgen E, Trautwein EA, Lapsley KG, Holmes C, Josse RG, Leiter LA, Connelly PW, Singer W. Assessment of the longer-term effects of a dietary portfolio of cholesterol-lowering foods in hypercholesterolemia. Am J Clin Nutr. 2006 Mar;83(3):582-91. doi: 10.1093/ajcn.83.3.582. PMID 16522904
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner D, Vidgen E, Lapsley KG, Trautwein EA, Parker TL, Josse RG, Leiter LA, Connelly PW. The effect of combining plant sterols, soy protein, viscous fibers, and almonds in treating hypercholesterolemia. Metabolism. 2003 Nov;52(11):1478-83. doi: 10.1016/s0026-0495(03)00260-9. PMID 14624410
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner DA, Wong JM, de Souza R, Emam A, Parker TL, Vidgen E, Lapsley KG, Trautwein EA, Josse RG, Leiter LA, Connelly PW. Effects of a dietary portfolio of cholesterol-lowering foods vs lovastatin on serum lipids and C-reactive protein. JAMA. 2003 Jul 23;290(4):502-10. doi: 10.1001/jama.290.4.502. PMID 12876093
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 Aug 21;8(8):CD011737. doi: 10.1002/14651858.CD011737.pub3. PMID 32827219
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 May 19;5(5):CD011737. doi: 10.1002/14651858.CD011737.pub2. PMID 32428300